CLINICAL TRIAL: NCT07055698
Title: Responsiveness And Minimal Clinically Important Difference Of Navicular Height Drop Test In Patients With Plantar Fasciitis
Brief Title: Responsiveness And Minimal Clinically Important Difference Of Navicular Height Drop Test With Plantar Fasciitis
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/832
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Navicular Height Drop (NHD) test — Evaluating the test's responsiveness and minimal clinically important difference (MCID) can help determine its clinical relevance in monitoring treatment outcomes.

SUMMARY:
Plantar fasciitis is a common musculoskeletal condition characterized by heel pain and impaired foot function, often linked to abnormal foot biomechanics. The Navicular Height Drop (NHD) test is a non-invasive tool used to assess dynamic foot posture by measuring changes in the medial longitudinal arch. Evaluating the test's responsiveness and minimal clinically important difference (MCID) can help determine its clinical relevance in monitoring treatment outcomes. Study objective to evaluate the responsiveness and determine the minimal clinically important difference (MCID) of the Navicular Height Drop (NHD) test in patients with plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of Plantar Fasciitis confirmed by Orthopedic presence of heel pain, particularly at the plantar aspect of the heel, for more than 3 months.
* Pain on palpation of the medial calcaneal tubercle.
* Positive Windlass test.
* Adults aged 25-60 years.
* Patients should be able to perform the Navicular Drop Test without any other concurrent - lower limb pathology that might interfere with the test (e.g., Achilles tendonitis, knee osteoarthritis, etc.).

Exclusion Criteria:

* Patients who have undergone any surgical intervention in the foot or ankle (e.g., plantar fascia release, foot fracture surgery).
* Recent history (within 6 weeks) of acute foot or ankle injury (e.g., fractures, sprains).
* Conditions such as rheumatoid arthritis, diabetes, neuropathy, peripheral vascular disease, or any neurological disorders affecting the lower limbs that could confound the results.
* Patients with other foot conditions like flatfoot deformity, bunion deformity, Morton's neuroma, severe hallux valgus, or any other condition affecting foot biomechanics that might alter the Navicular Drop Test results.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A Perspective Cohort Study. This study aims to establish the responsiveness and MCID of the NHD test, enabling its effective use as a clinical tool for monitoring plantar fasciitis outcomes. By identifying clinically meaningful changes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Navicular Height Drop Test (NHDT) | 12 Months
  This test measures the change in the position of the navicular bone during weight-bearing, helping to assess foot arch collapse and the impact of abnormal foot biomechanics, which is crucial in conditions like plantar fasciitis
GLOBAL RATING OF CHANGE (GRC) | 12 Months
  The GRC scale is a simple tool where patients rate their overall improvement after treatment. It is often used to establish the MCID by comparing patients' subjective perceptions of improvement with changes in objective measures like NHDT. The responses are usually rated on a Likert-type scale, which might look like this:+7: Very Much Improved ,+6: Much Improved ,+5: Improved ,+4: Minimally Improved ,+3: No Change ,+2: Minimally Worse ,+1: Worse ,0: Very Much Worse(31).
Foot Function Index | 12 Months
  A self-reported questionnaire assessing pain, disability, and activity limitation in individuals with foot disorders, commonly used to assess the functional impact of plantar fasciitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Omer Hospital & Cardiac Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No